CLINICAL TRIAL: NCT05079191
Title: Diagnostic Performance and Predictive Impact of the CT Scan in Patients With Suspected Covid-19
Brief Title: Impact of the CT Scan in Patients With Suspected Covid-19
Acronym: SCAN-COV-HUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7844
Record Dates: First submitted 2021-10-14; First posted 2021-10-15 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; Chest scanner; CT scan; RT-PCR
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnostic performance of the scanner in the indication of suspected Covid-19 is not yet well known, especially in comparison with the results of RT-PCR.

The potential use of the scanner as a tool for quantifying the severity of Covid-19 disease is not yet well established, especially the variations between readers or between measurement techniques.

The impact of the scanner in predicting the fate of patients with confirmed Covid-19 is not yet known.

ELIGIBILITY:
Inclusion criteria

* Adult patient (≥18 years old)
* Patient admitted to Strasbourg University Hospitals for suspicion of Covid-19, between 03/01/2020 and 04/29/2020
* Availability of at least one chest CT scan during hospitalization
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Non-inclusion criteria

* Patient who expressed his opposition to participating in the study
* Patient under legal protection
* Patient under guardianship or guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient admitted to Strasbourg University Hospitals for suspicion of Covid-19
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the chest scanner in suspected Covid-19 | Files analysed retrospectively from March 01, 2020 to April 29, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie B - Hôpitaux Universitaires de Strasbourg, Strasbourg, France